CLINICAL TRIAL: NCT01724892
Title: Comparison the Effects of Dexamethasone and Loteprednol on Epithelial Healing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Onsiri Thanathanee, othana, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: othana001
Record Dates: First submitted 2012-11-06; First posted 2012-11-12 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Epithelial Defect After Phototherapeutic Keratectomy
MeSH Terms: interventions — Dexamethasone; Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loteprednol etabonate (Active Comparator): Topical Loteprednol etabonate eye drop 0.5%, 4 times a day, 3 weeks
  Interventions: Drug: Dexamethasone
- Dexamethasone (Active Comparator): Topical Dexamethasone eye drop 0.1%, 4 times a day, 3 weeks
  Interventions: Drug: Loteprednol etabonate

INTERVENTIONS:
Drug: Dexamethasone
  Arms: Loteprednol etabonate
Drug: Loteprednol etabonate
  Arms: Dexamethasone

SUMMARY:
Corticosteroid has been used for the treatment after phototherapeutic keratectomy (PRK). Dexamethasone, a potent steroid can retard the corneal epithelial healing rate and has numerous serious complications, especially glaucoma. Loteprednol, a new generation of corticosteroid has less potency than dexamethasone and was proposed to has less side effect regarding intraocular pressure (IOP) elevation. Therefore, Investigators would like to compare the effect of dexamethasone and loteprednol on corneal epithelial healing rate after PRK and risk of glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* the patient with epithelial defect after phototherapeutic keratectomy

Exclusion Criteria:

* the patient with systemic disease such as diabetes and connective tissue disease
* the patient with ocular surface disease such as dry eye and recurrent corneal erosion

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
corneal epithelial healing | 1 month

SECONDARY OUTCOMES:
intraocular pressure | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Onsiri Thanathanee, MD, Principal Investigator — Khon Kaen University
Locations (2):
- Thailand (2):
  - Onsiri Thanathanee, Khon Kaen, Changwat Khon Kaen
  - Srinagarind Hospital, Khon Kaen, Changwat Khon Kaen

REFERENCES:
- [Background] Amon M, Busin M. Loteprednol etabonate ophthalmic suspension 0.5 %: efficacy and safety for postoperative anti-inflammatory use. Int Ophthalmol. 2012 Oct;32(5):507-17. doi: 10.1007/s10792-012-9589-2. Epub 2012 Jun 16. PMID 22707339
- [Derived] Thanathanee O, Sriphon P, Anutarapongpan O, Athikulwongse R, Thongphiew P, Rangsin R, Suwan-apichon O. A randomized controlled trial comparing dexamethasone with loteprednol etabonate on postoperative photorefractive keratectomy. J Ocul Pharmacol Ther. 2015 Apr;31(3):165-8. doi: 10.1089/jop.2014.0107. Epub 2015 Jan 2. PMID 25555173
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed?term=dexamethasone%20AND%20loteprednol